CLINICAL TRIAL: NCT05831228
Title: Effects of Pre-dive Ketone Food Products on Latency to Central Nervous System Oxygen Toxicity
Brief Title: Effects of Pre-dive Ketone Food Products on Latency to CNS Oxygen Toxicity (Aim 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Navy (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00111000_1
Record Dates: First submitted 2023-03-24; First posted 2023-04-26 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Oxygen Toxicity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Ketogenic food products (Experimental): Dietary Supplement: Ketogenic food products Participants will be given a ketogenic food product prior to the hyperbaric oxygen exposure.
  Interventions: Dietary Supplement: Ketogenic food products
- Control: Placebo (Placebo Comparator): Dietary Supplement comparator
  Interventions: Dietary Supplement: Control: Placebo

INTERVENTIONS:
Dietary Supplement: Ketogenic food products — Participants will be given a ketogenic food product prior to the hyperbaric oxygen exposure.
  Arms: Experimental: Ketogenic food products
Dietary Supplement: Control: Placebo — Participants will be given a dietary supplement comparator prior to the hyperbaric oxygen exposure.
  Arms: Control: Placebo

SUMMARY:
The purpose of this study is to understand how ketogenic food products affect oxygen toxicity in undersea divers. Oxygen toxicity affecting the central nervous system, mainly the brain, is a result of breathing higher than normal oxygen levels at elevated pressures as can be seen in SCUBA diving or inside a hyperbaric (pressure) chamber. This is a condition that may cause a wide variety of symptoms such as: vision disturbances, ear-ringing, nausea, twitching, irritability, dizziness, and potentially loss of consciousness or seizure. Because nutritional ketosis has been used to reduce or eliminate seizures in humans, it may be beneficial to reduce oxygen toxicity as well. The investigators hope this study will provide a help to develop practical and useful methods for improving the safety of undersea Navy divers, warfighters and submariners.

DETAILED DESCRIPTION:
Central nervous system (CNS) oxygen toxicity continues to be a risk for military divers and constrains their operations. Manifestations of this condition range from nausea, twitching, and tinnitus to seizures and unresponsiveness, and the latter may lead to death by drowning. The NAVY has a need for better methods to prevent or delay the onset of CNS oxygen toxicity (CNSOT) and to safely expand the scope of diving operations. It is the broad objective of this study to generate information that will enhance warfighter safety and performance in relevant NAVY operations by reducing the risk of CNS oxygen toxicity.

It is known that nutritional ketosis through a diet with a high fat-to-carbohydrate ratio (ketogenic diet) can reduce the frequency and severity of epileptic seizures in humans, and a recent animal study has shown that dietary ketosis also delays the onset of CNSOT. In recent years, ketone ester food products ketone esters have been made commercially available which may elevate circulating ketone levels. The investigators aim to investigate whether ketosis from commercially available ketogenic food products prior to a dive will delay the onset of CNSOT.

The first aim of this study will be to determine the effect of ketone food product ingestion on serum ketone levels, and document any relevant side effects. Post-ingestion ketone levels will be trended for 3 different ketone food product regimens in 15 total subjects. Data will be used to select the optimal ketone food product strategy to investigate in the second aim.

This second aim will be to evaluate the primary hypothesis, that pre-dive ketone food products will prolong latency to CNSOT. To assess this, 20 subjects will be studied in a randomized, controlled, double-blind, crossover methodology. After consuming either the ketone food product or placebo, each subject will complete an immersed, head out hyperbaric oxygen exposure while exercising on an underwater cycle ergometer at 2.06 ATA (35 fsw) until oxygen toxicity symptoms develop or the maximum time limit of 120 minutes is reached. The experiment will be repeated on a different day by each subject after consuming the opposite (ketone food products or placebo). Primary outcome will be time to manifestation of CNSOT. Physiologic monitoring throughout the study will provide secondary endpoints such as cognitive performance, sympathetic nervous system stimulation via electrodermal activity, electroencephalography, cardiorespiratory measures and end-tidal CO2/O2/N2; all adding to our understanding of CNSOT physiology which may guide future mitigation and monitoring strategies.

ELIGIBILITY:
Inclusion Criteria:

* Males & females between 18 and 39 years old.
* Measured (Phase 2) VO2max ≥ 30 ml/kg/min (female) or 35 ml/kg/min (male).
* BMI ≤ 30.0 unless VO2max and baseline exercise profile is deemed appropriate for the study by the PI.
* (Phase 2 only) Able to exercise continuously on cycle ergometer for 2 hours.
* (Phase 2 only) Able to equalize middle ears and tolerate hyperbaric chamber exposure test.

Exclusion Criteria:

* Prolonged QTc on initial ECG
* Currently pregnant or attempting to become pregnant.
* Have a medical history of:

  1. Smoking history deemed significant by PI
  2. Known significant electrolyte disorders
  3. Coronary artery disease
  4. Cardiac arrhythmia deemed significant by PI
  5. Lung disease
  6. Hypertension
  7. Seizures
  8. Exercise intolerance or inability to meet inclusion requirements
  9. Psychiatric disorder deemed significant by PI
  10. Previous pneumothorax or pneumomediastinum
  11. Hypo- or hyperglycemia
  12. Diabetes
  13. Inability to equalize middle ear spaces during hyperbaric compression
  14. Claustrophobia
* Regularly take any medications which may alter heart rate, blood pressure, neurotransmitter function, alter seizure threshold, mood or affect per PI discretion.
* Any other condition limiting ability to perform exercise testing or dive profile as determined by the investigators.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Latency to central nervous system oxygen toxicity (CNSOT) | 2 hours
  Assessment of latency to CNSOT in a simulated working dive breathing 100% oxygen at 2.06 ATA, immersed in water (head out), in a hyperbaric chamber while performing exercise. Endpoint is time to development of signs or symptoms of CNSOT. Maximum duration 120 minutes.

SECONDARY OUTCOMES:
Cognitive performance | Day 1
  Changes in Multi Attribute Test battery scores prior to and during hyperbaric exposure. Tracking score pixel distance from target center, scale min = 0, no defined maximum.
Level of nutritional ketosis as detected by serume beta hydroxybutyrate levels | Day 1
  Measure serume beta hydroxybutyrate levels in blood samples
Number of participants with change in EEG | Day 1
  Changes in visual EEG inspection prior to and during hyperbaric exposure.
Change in qEEG alpha/delta power ratio (ratio of power in alpha frequency band to power in delta frequency band) | Day 1
  Changes in qEEG readings prior to and during hyperbaric exposure
Change in end-tidal CO2 | Day 1
  Changes in end-tidal CO2 levels in blood samples prior to and during hyperbaric exposure
Change in venous CO2 | Day 1
  Changes in CO2 levels in blood samples prior to and during hyperbaric exposure
Change in heart rate | Day 1
  Changes in heart rate prior to and during hyperbaric exposure
Change in ventilatory rate | Day 1
  Changes in ventilatory rate prior to and during hyperbaric exposure
Number of participants who develop CNS oxygen toxicity | Day 1
  Any symptoms of CNSOT during hyperbaric exposure as described by participants will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Derrick, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT05831228/ICF_000.pdf